CLINICAL TRIAL: NCT03022552
Title: Heart Attack Research Program: Platelet Sub-Study (HARP); Platelet Collection for Patients With Myocardial Infarction
Brief Title: Heart Attack Research Program: Platelet Sub-Study (HARP)
Acronym: HARP
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 16-01104-3
Record Dates: First submitted 2017-01-13; First posted 2017-01-16 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; Platelets; Blood Collection; Genomics
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood Collection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MINOCA: Women with myocardial infarction (MI) with demonstrated non-obstructive coronary artery disease during cardiac catheterization (less than 50% blockage in any major vessel).
- MI-CAD: Women with myocardial infarction (MI) with demonstrated obstructive coronary artery disease during cardiac catheterization (50% or greater blockage in any major vessel) or previous history of percutaneous coronary intervention (PCI) or or coronary artery bypass graft (CABG).
- CATH-NOCA: Women with stable angina that are age and race matched to women in the MINOCA arm that are clinically referred for cardiac catheterization

SUMMARY:
This prospective observational cohort study, will investigate the platelet phenotype, platelet genetic composition, and role of platelets as effector cells in women and men with myocardial infarction (MINOCA or MI-CAD) and controls. This study, which will take place at NYU and Bellevue Medical Center, and participating external sites. May have concurrent enrollment with the HARP Main Imaging (NCT02914483). Additionally, a sex, group of age and race matched disease controls 'CATH-NOCA' composed of women and men with stable angina referred for cardiac catheterization, will be enrolled. Blood obtained during the initial catheterization and 2 months post-MI will be utilized for platelet testing.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic symptoms compatible with diagnosis of MI, such as chest pain or anginal equivalent symptoms at rest or new onset exertional anginal equivalent symptoms
* Objective evidence of MI (either or both of the following):

  * Elevation of troponin to above the laboratory upper limit of normal (ULN)
  * ST segment elevation of ≥1mm on 2 contiguous ECG leads
* Willing to provide informed consent and comply with all aspects of the protocol
* Administration of aspirin at least 1 hour before cardiac catheterization
* Administration of thienopyridine (e.g., clopidogrel, ticagrelor) at least 1 hour before cardiac catheterization
* Women and men with ≥50% of any major epicardial vessel on invasive angiography may participate

Exclusion Criteria:

* Recent use of vasospastic agents, such as cocaine, triptans, or ergot alkaloids (≤1 month)
* Alternate explanation for troponin elevation, such as hypertensive urgency, acute exacerbation of heart failure, chronic elevation due to kidney disease, pulmonary embolism, cardiac trauma
* Pregnancy
* Thrombolytic therapy for STEMI (qualifying event)
* Use of any of the following medications:
* Platelet antagonists (except aspirin and thienopyridines) within 7 days
* NSAIDs (e.g., ibuprofen, naproxen) within 3 days.
* Thrombocytopenia (platelet count <100,000)
* Thrombocytosis (platelet count >500,000)
* Anemia (hemoglobin <9 mg/dl)
* Hemorrhagic diathesis

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study may have concurrent enrollment with the HARP Main Imaging (NCT02905357). This study population includes women and men who present to the hospital with an MI, with non-obstructive coronary artery disease or obstructive artery disease, are eligible for blood collection. Additionally, a sex, group of age and race matched disease controls 'CATH-NOCA' will be composed of women and men with stable angina referred for cardiac catheterization.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Examination of Platelet Activity Markers | 1 year
Examination of Markers of Cardiovascular Disease Risk | 1 year
  This will include additional examination of known thrombosis, Inflammation, metabolic disease, and lipids/lipoprotein markers.
Cellular and molecular mechanism of myocardial infarction in women | 1 year
  To further investigate this mechanism, recent advances in microRNA, RNA, DNA expression profiling, and plasma and serum collections will be used.

SECONDARY OUTCOMES:
Examination of non-coding and coding mRNA profiles in women with MI and matched controls | 4 years
  Specific transcripts associated with platelet activation, plaque destabilization, and different cardiovascular diseases will be analyzed at the genetic level.

CONTACTS AND LOCATIONS:
Overall Officials: Harmony R Reynolds, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared after the end of the study.

REFERENCES:
- [Derived] Sowa MA, Hannemann C, Pinos I, Ferreira E, Biwas B, Dai M, Corr EM, Cornwell MG, Drenkova K, Lee AH, Spruill T, Reynolds HR, Hochman JS, Ruggles KV, Campbell RA, van Solingen C, Wright MD, Moore KJ, Berger JS, Barrett TJ. Tetraspanin CD37 regulates platelet hyperreactivity and thrombosis. Cardiovasc Res. 2025 Jun 12;121(6):943-956. doi: 10.1093/cvr/cvaf051. PMID 40126944
- [Derived] Barrett TJ, Corr EM, van Solingen C, Schlamp F, Brown EJ, Koelwyn GJ, Lee AH, Shanley LC, Spruill TM, Bozal F, de Jong A, Newman AAC, Drenkova K, Silvestro M, Ramkhelawon B, Reynolds HR, Hochman JS, Nahrendorf M, Swirski FK, Fisher EA, Berger JS, Moore KJ. Chronic stress primes innate immune responses in mice and humans. Cell Rep. 2021 Sep 7;36(10):109595. doi: 10.1016/j.celrep.2021.109595. PMID 34496250
- [Derived] Barrett TJ, Lee AH, Smilowitz NR, Hausvater A, Fishman GI, Hochman JS, Reynolds HR, Berger JS. Whole-Blood Transcriptome Profiling Identifies Women With Myocardial Infarction With Nonobstructive Coronary Artery Disease. Circ Genom Precis Med. 2018 Dec;11(12):e002387. doi: 10.1161/CIRCGEN.118.002387. No abstract available. PMID 30562118